CLINICAL TRIAL: NCT04930744
Title: A Prospective, Randomized Open-Label Phase II Study of the Safety and Tolerability of Metformin in Combination With Standard Antimicrobial Treatment of Pulmonary Tuberculosis in People With TB and Co-infected With HIV
Brief Title: Safety and Tolerability of Metformin in People With Tuberculosis (TB) and Human Immunodeficiency Virus (HIV)
Acronym: METHOD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Aurum Institute (Other); A*STAR Infectious Diseases Labs (Industry); University of Cape Town (Other); Wits Health Consortium (Pty) Ltd (Other)
Responsible Party: Principal Investigator, Hardy Kornfeld, MD, Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AUR1-1-199; 5U01AI134585 (NIH)
Record Dates: First submitted 2021-05-26; First posted 2021-06-18 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Tuberculosis; Pulmonary Tuberculosis; HIV Coinfection
Keywords: Metformin; Tuberculosis; Anti-Tuberculosis Treatment (ATT); Anti-Viral Therapy (ART)
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary; HIV Infections | interventions — Isoniazid; Rifampin; Ethambutol; Pyrazinamide; Metformin

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two or more groups, Standard ATT or Standard ATT plus Metformin in parallel for 11 weeks starting 1 week after ATT initiation.
Masking Description: Senior study leadership, Drs. Kornfeld, Wallis, Churchyard, Singhal will be blinded. Participants, study personnel and clinicians are not blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard Tuberculosis Medicine (Active Comparator): Participants will have a chance to be put on standard tuberculosis medicines (Isoniazid, Rifampicin, Ethambutol and Pyrazinamide) only. It is a combination pill pack that will be taken by mouth daily. The combination pack includes Isoniazid, Rifampicin, Ethambutol, and Pyrazinamide which they will take for 2 months. They will only take Isoniazid and Rifampicin for the last 4 months.
  Interventions: Drug: Isoniazid; Drug: Rifampicin; Drug: Ethambutol; Drug: Pyrazinamide
- Standard TB Medicines and Metformin (Experimental): Participants will have a chance to be put on standard tuberculosis medicines (Isoniazid, Rifampicin, Ethambutol and Pyrazinamide) only. It is a combination pill pack that will be taken by mouth daily. The combination pack includes Isoniazid, Rifampicin, Ethambutol, and Pyrazinamide which they will take for 2 months. They will only take Isoniazid and Rifampicin for the last 4 months. For this arm, they will also take Metformin hydrochloride one 500 mg tablet daily starting one week after the initiation of tuberculosis medicines, then increasing to one 500 mg table twice daily through study week-12 for a total 11 weeks of metformin exposure.
  Interventions: Drug: Isoniazid; Drug: Rifampicin; Drug: Ethambutol; Drug: Pyrazinamide; Drug: Metformin hydrochoride

INTERVENTIONS:
Drug: Isoniazid — Isoniazid, dose prescribed by participant's physician, will be taken by mouth daily. Isoniazid, is in a combination pill pack with the other standard ATT medications.
Drug: Rifampicin — Rifampicin, dose prescribed by participant's physician, will be taken by mouth daily. Rifampicin is in a combination pill pack with the other standard ATT medications.
Drug: Ethambutol — Ethambutol, dose prescribed by participant's physician, will be taken by mouth daily. Ethambutol is in a combination pill pack with the other standard ATT medications.
  Other Names: Myambutol
Drug: Pyrazinamide — Pyrazinamide, dose prescribed by participant's physician, will be taken by mouth daily. Pyrazinamide is in a combination pill pack with the other standard ATT medications.
Drug: Metformin hydrochoride — Metformin hydrochloride 500 mg tablet once daily starting one week after the initiation of TB treatment, then increasing to study twice daily through study week-12 (11 weeks total metformin treatment).
  Other Names: Glucophage
  Arms: Standard TB Medicines and Metformin

SUMMARY:
The METHOD study will examine whether adding metformin to standard antibiotic treatment for tuberculosis (TB) in people with HIV is safe and well tolerated. The study will also test if adding metformin clears the infection more quickly and with less lung damage. When enrolled, participants will have an equal chance of being in the group that takes standard TB medicines alone or in the group that also takes metformin. Participants will have a chance to be put on either: 1) standard TB medicines (isoniazid, rifampicin, ethambutol and pyrazinamide for two months, continuing isoniazid and rifampin for four more months) only; or 2) the same standard TB medicines plus metformin. Participants randomized to the metformin arm will take metformin for eleven weeks, starting one week after starting the standard TB medicines. In addition to monitoring for side effects, all participants will have studies of drug levels and lung and immune function.

DETAILED DESCRIPTION:
The METHOD trial is a Phase II A randomized, open-label trial of metformin added to standard anti-tuberculosis treatment (ATT) and anti-retroviral therapy (ART) in TB/HIV co-infected patients. HIV-positive adults (treated or ART-naïve) newly diagnosed with sputum culture-positive, drug-sensitive pulmonary TB will be recruited to and enrolled in the study. All participants in the interventional study will take standard ATT for drug-sensitive pulmonary TB starting at enrollment. Participants in the metformin arm will begin taking metformin 1 week later and metformin will be stopped on week-12. The "omics" control group will include those (treated or ART-naïve) without evidence of active TB. The total cohort is sample size N=112, comprising 56 participants each in two parallel study arms (standard therapy or standard therapy plus metformin) with the goal of retaining 100 participants with evaluable data for analysis. The duration of the METHOD trial is 5 years. The duration of individual participation in the interventional arms of the study is 36 weeks, not including an initial period of screening over an interval of up to 14 additional days prior to study enrollment. The final clinic visit coincides with the completion of ATT at week-24. The final follow-up contact is a phone interview at week-36. Ten consenting participants from each study arm (n=20 total) will have intensive pharmacokinetic/pharmacodynamic (PK/PD) sampling. The remaining 92 participants will have sparse PK/PD sampling.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 through 65 years.
2. HIV-1 seropositive status prior to or after screening.
3. Chest radiograph compatible with pulmonary TB.
4. Positive sputum Xpert TB/RIF or Ultra with one CT <25.
5. RIF susceptibility diagnosed by Xpert TB/RIF or Ultra.
6. Residence within study catchment area.
7. If female of childbearing potential, willing to use contraception for the duration of study participation (Criteria for childbearing potential and for acceptable contraception). If male, willing to use condoms for the duration of metformin treatment plus 3 months after stopping metformin.
8. Able and willing to provide informed consent. Inclusion criteria 1, 2, 6, 7, and 8 also apply to the control group.

Exclusion criteria:

1. Any condition for which participation in the trial, as judged by the investigator, could compromise the well-being of the subject or prevent, limit or confound protocol-specified assessments.
2. Is critically ill, and in the judgment of the investigator has a diagnosis likely to result in death during the trial or the follow-up period.
3. TB meningitis or other forms of severe TB with high risk of a poor outcome as judged by the investigator.
4. Pregnant or breastfeeding.
5. Resistance to any first-line ATTB drug demonstrated by susceptibility testing.
6. More than 14 days ATT for the current episode of TB, prior to enrollment.
7. Taking any fluoroquinolone antibiotic.
8. History of diabetes mellitus or fasting blood glucose >7.0 mmol/L on screening evaluation
9. History of congestive heart failure, chronic liver disease, diabetes, autoimmune disease or malignancy.
10. Consumption of >28 units (men) OR >21 units (women) of alcohol/week (see Protocol Appendix; Alcohol Pre-Screening Checklist).
11. Use of metformin within 1 year prior to enrollment.
12. History of sensitivity to metformin.
13. Acute or chronic metabolic acidosis based on reported medical history or laboratory tests performed on screening.
14. Body mass index (BMI) <17.0 kg/m2 on screening evaluation.
15. Peripheral blood CD4 T cell count <50 cells/mm3 on screening evaluation.
16. Hemoglobin <9 g/dL for males, and <8 g/dL (women) for females on screening evaluation.
17. Platelet count <50,000/mm3 on screening evaluation.
18. Absolute neutrophil count <750 cells/mm3 on screening evaluation.
19. Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m2 calculated by the CKD-EPI equation.
20. Serum bicarbonate <18 mmol/L on screening evaluation.
21. AST or ALT ≥3 times the upper limit of normal (ULN) on screening evaluation.
22. Hepatitis B surface antigen positive.
23. Enrollment in another interventional study at any time during participation in the METHOD trial.
24. Imprisonment at the time of or after enrollment in the METHOD trial.
25. Diagnosis of active COVID-19 at the time of screening or high suspicion of active COVID-19 disease during screening.

Exclusion criteria 1, 2, 4, 5, 7, 8-11, 13-25 also apply to participants in the omics control group. In addition, a positive sputum Xpert TB/RI, Mtb culture or any radiographic evidence of any pulmonary infectious disease process is exclusion criteria for the omics control group.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity.
Enrollment: 112 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2025-04-19 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of metformin as measured by the number of grade 3 or higher gastrointestinal (GI) adverse events | Up to 16 weeks
  Average and median numbers of Grade 3, 4 and 5 adverse events will be tabulated by treatment arm

SECONDARY OUTCOMES:
Metformin added to standard ATT improves respiratory health as measured by radiographic score | Change in baseline radiographic score at week 24
  Between arm differences of change in radiographic score will be tabulated by arm and time point.
Metformin added to standard ATT improves respiratory health as measured by 6-minute Walk Test (6MWT) as assessed by distance x 02 saturation (2° endpoint) | Change in baseline 6MWT at week 24
  Between arm differences of change in 6MWT distance oxygen saturation will be tabulated by arm and time point.
Metformin added to standard ATT improves respiratory health as measured by spirometry: Forced Vital Capacity (FVC) | Change in baseline spirometric value at week 24
  Between arm differences of change in spirometric values will be tabulated by arm and time point.
Metformin added to standard ATT improves respiratory health as measured by spirometry: Forced Expiratory Volume (FEV1%) (2° endpoint) | Change in baseline spirometric value at week 24
  Between arm differences of change in spirometric values will be tabulated by arm and time point.
Metformin added to standard ATT improves respiratory health as measured by Saint George's Respiratory Questionnaire (SGRQ) assessed by 2° endpoint | Change in baseline SGRQ at week 24
  Between arm differences of change in SGRQ score will be tabulated by arm and timepoint.
Metformin added to standard ATT improves HIV outcomes as measured by HIV viral load | Up to 24 weeks
  Between-arm differences of HIV viral load
Metformin added to standard ATT improves HIV outcomes as measured by CD4 | Up to 24 weeks
  Between-arm differences in CD4
Metformin added to standard ATT improves HIV outcomes as measured by T cell count | Up to 24 weeks
  Between-arm differences of T cell count
Metformin added to standard ATT improves TB treatment outcomes | Up to 24 weeks
  Between arm differences will be tabulated in the secondary endpoints of cure, failure, death, default, and relapse.

OTHER OUTCOMES:
Efficacy of metformin as measured by time to sputum conversion in Mycobacterial Growth Indicator Tube (MGIT) | Up to 24 weeks
  Sputum liquid culture conversion will be tabulated by treatment arm

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Wallis, MD, FIDSA, Study Chair — Aurum Institute; Hardy Kornfeld, MD, Principal Investigator — The University of Massachusetts Chan Medical School
Locations (2):
- South Africa (2):
  - Tembisa Clinical Research Centre-The Aurum Institute, Johannesburg, Gauteng
  - Isango Lethemba TB Research Unit, Port Elizabeth

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share the standard operating procedures, the study protocol, the informed consent form, and the data collection tools. Research data that document, support and validate research findings will be made available after the main findings from the final research data set have been accepted for publication. The trial also includes a plan to collect and store genomic DNA. Written informed consent is obtained indicating consent for their genomic and phenotypic data to be used for future research purposes and to be shared broadly in a de-identified manner. Institutional certification has been obtained. Data generated from this trial, including genomic data and associated data, will be submitted to an NIH-designated repository such as database of Genotype and Phenotype (dbGaP).
Supporting Information: Study Protocol, ICF
Time Frame: Data generated by this investigation will be made publicly available no later than six months after the initial data submission to NIH or at the time of the first publication, whichever occurs first.
Access Criteria: Following publication of research data, may be shared upon request by contacting the study principal investigators by email.

REFERENCES:
- [Background] Divecha N, Mansouri H, Peat D, Cope G, Partridge L, McDonald CJ. Isoprenaline-induced and constitutive members of a proline-rich protein sub-group from mouse parotid glands studied with monoclonal antibody NAL1. J Mol Endocrinol. 1989 Jul;3(1):7-14. doi: 10.1677/jme.0.0030007. PMID 2742745
- [Background] Chap Z, Ishida T, Jones RH, Pena JR, Vinik A, Field JB. Hepatic extraction of somatostatin in conscious dogs. Am J Physiol. 1988 Feb;254(2 Pt 1):E214-21. doi: 10.1152/ajpendo.1988.254.2.E214. PMID 2894771
- [Background] Shperling ID. [A rare case of implantation metastases of a melanoma to the mitral valve with embolism of the coronary artery, infarct and myocardial rupture]. Arkh Patol. 1989;51(6):70-2. Russian. PMID 2803032
- [Background] Singhal A, Jie L, Kumar P, Hong GS, Leow MK, Paleja B, Tsenova L, Kurepina N, Chen J, Zolezzi F, Kreiswirth B, Poidinger M, Chee C, Kaplan G, Wang YT, De Libero G. Metformin as adjunct antituberculosis therapy. Sci Transl Med. 2014 Nov 19;6(263):263ra159. doi: 10.1126/scitranslmed.3009885. PMID 25411472
- [Background] Strate SM, Rutledge JC, Weinberg AG. Delayed development of angiosarcoma in multinodular infantile hepatic hemangioendothelioma. Arch Pathol Lab Med. 1984 Dec;108(12):943-4. No abstract available. PMID 6548897
- [Background] Dubarry JJ, Auche Y, Bernard JP, Fontanges X. [Therapeutic application of anabolising drugs in gastroenterology. Apropos of Primobolan-Depot]. Gaz Med Fr. 1965 Sep 10;72(17):2896-8. No abstract available. French. PMID 5848303
- [Background] Kumar NP, Moideen K, Viswanathan V, Shruthi BS, Sivakumar S, Menon PA, Kornfeld H, Babu S. Elevated levels of matrix metalloproteinases reflect severity and extent of disease in tuberculosis-diabetes co-morbidity and are predominantly reversed following standard anti-tuberculosis or metformin treatment. BMC Infect Dis. 2018 Jul 25;18(1):345. doi: 10.1186/s12879-018-3246-y. PMID 30045688
- [Background] Padmapriyadarsini C, Bhavani PK, Natrajan M, Ponnuraja C, Kumar H, Gomathy SN, Guleria R, Jawahar SM, Singh M, Balganesh T, Swaminathan S. Evaluation of metformin in combination with rifampicin containing antituberculosis therapy in patients with new, smear-positive pulmonary tuberculosis (METRIF): study protocol for a randomised clinical trial. BMJ Open. 2019 Mar 1;9(3):e024363. doi: 10.1136/bmjopen-2018-024363. PMID 30826761
- [Background] Bianchi Porro G, Parente F. Recent developments in peptic ulcer treatment. Scand J Gastroenterol Suppl. 1988;146:159-65. doi: 10.3109/00365528809099142. PMID 2906460
- [Background] Vincenzoni M, Brizi MG, De Vivo D, Romani M, Del Grosso C, Vecchioli A. Computerised management of the radio-diagnostic ward: considerations on our three years experience. Rays. 1985 May-Aug;10(2):57-61. No abstract available. PMID 3843655
- [Background] Ralph AP, Ardian M, Wiguna A, Maguire GP, Becker NG, Drogumuller G, Wilks MJ, Waramori G, Tjitra E, Sandjaja, Kenagalem E, Pontororing GJ, Anstey NM, Kelly PM. A simple, valid, numerical score for grading chest x-ray severity in adult smear-positive pulmonary tuberculosis. Thorax. 2010 Oct;65(10):863-9. doi: 10.1136/thx.2010.136242. PMID 20861290
- [Background] Salpeter SR, Greyber E, Pasternak GA, Salpeter EE. Risk of fatal and nonfatal lactic acidosis with metformin use in type 2 diabetes mellitus. Cochrane Database Syst Rev. 2010 Apr 14;2010(4):CD002967. doi: 10.1002/14651858.CD002967.pub4. PMID 20393934
- [Background] Graham GG, Punt J, Arora M, Day RO, Doogue MP, Duong JK, Furlong TJ, Greenfield JR, Greenup LC, Kirkpatrick CM, Ray JE, Timmins P, Williams KM. Clinical pharmacokinetics of metformin. Clin Pharmacokinet. 2011 Feb;50(2):81-98. doi: 10.2165/11534750-000000000-00000. PMID 21241070
- [Background] Chandel NS, Avizonis D, Reczek CR, Weinberg SE, Menz S, Neuhaus R, Christian S, Haegebarth A, Algire C, Pollak M. Are Metformin Doses Used in Murine Cancer Models Clinically Relevant? Cell Metab. 2016 Apr 12;23(4):569-70. doi: 10.1016/j.cmet.2016.03.010. No abstract available. PMID 27076070
- [Background] Song IH, Zong J, Borland J, Jerva F, Wynne B, Zamek-Gliszczynski MJ, Humphreys JE, Bowers GD, Choukour M. The Effect of Dolutegravir on the Pharmacokinetics of Metformin in Healthy Subjects. J Acquir Immune Defic Syndr. 2016 Aug 1;72(4):400-7. doi: 10.1097/QAI.0000000000000983. PMID 26974526
- [Background] Te Brake LHM, Yunivita V, Livia R, Soetedjo N, van Ewijk-Beneken Kolmer E, Koenderink JB, Burger DM, Santoso P, van Crevel R, Alisjahbana B, Aarnoutse RE, Ruslami R; TANDEM Consortium. Rifampicin Alters Metformin Plasma Exposure but Not Blood Glucose Levels in Diabetic Tuberculosis Patients. Clin Pharmacol Ther. 2019 Mar;105(3):730-737. doi: 10.1002/cpt.1232. Epub 2018 Oct 29. PMID 30222857
- [Background] Allard M. My solidarity towards patients. Interview by Guylaine Campion. Infirm Aux. 1985 Oct;58(2):15-6, 32-3. No abstract available. English, French. PMID 3853537
- [Background] Wulffele MG, Kooy A, Lehert P, Bets D, Ogterop JC, Borger van der Burg B, Donker AJ, Stehouwer CD. Effects of short-term treatment with metformin on serum concentrations of homocysteine, folate and vitamin B12 in type 2 diabetes mellitus: a randomized, placebo-controlled trial. J Intern Med. 2003 Nov;254(5):455-63. doi: 10.1046/j.1365-2796.2003.01213.x. PMID 14535967
- [Background] Lalau JD. Lactic acidosis induced by metformin: incidence, management and prevention. Drug Saf. 2010 Sep 1;33(9):727-40. doi: 10.2165/11536790-000000000-00000. PMID 20701406
- [Background] Booysen HL, Woodiwiss AJ, Raymond A, Sareli P, Hsu HC, Dessein PH, Norton GR. Chronic kidney disease epidemiology collaboration-derived glomerular filtration rate performs better at detecting preclinical end-organ changes than alternative equations in black Africans. J Hypertens. 2016 Jun;34(6):1178-85. doi: 10.1097/HJH.0000000000000924. PMID 27035736
- [Background] DeFronzo R, Fleming GA, Chen K, Bicsak TA. Metformin-associated lactic acidosis: Current perspectives on causes and risk. Metabolism. 2016 Feb;65(2):20-9. doi: 10.1016/j.metabol.2015.10.014. Epub 2015 Oct 9. PMID 26773926
- [Background] Brackett CC. Clarifying metformin's role and risks in liver dysfunction. J Am Pharm Assoc (2003). 2010 May-Jun;50(3):407-10. doi: 10.1331/JAPhA.2010.08090. PMID 20452916
- [Background] Wallis RS, Peppard T. Early Biomarkers and Regulatory Innovation in Multidrug-Resistant Tuberculosis. Clin Infect Dis. 2015 Oct 15;61Suppl 3:S160-3. doi: 10.1093/cid/civ612. PMID 26409278
- [Background] Hoft DF, Worku S, Kampmann B, Whalen CC, Ellner JJ, Hirsch CS, Brown RB, Larkin R, Li Q, Yun H, Silver RF. Investigation of the relationships between immune-mediated inhibition of mycobacterial growth and other potential surrogate markers of protective Mycobacterium tuberculosis immunity. J Infect Dis. 2002 Nov 15;186(10):1448-57. doi: 10.1086/344359. Epub 2002 Oct 23. PMID 12404160
- [Background] Bone LB, Johnson KD. Treatment of tibial fractures by reaming and intramedullary nailing. J Bone Joint Surg Am. 1986 Jul;68(6):877-87. PMID 3733776
- [Background] Kosinska M. [Nursing decisions--their scope and limitations]. Pieleg Polozna. 1988;(4):6-7. No abstract available. Polish. PMID 3399551
- [Background] Aperis G, Paliouras C, Zervos A, Arvanitis A, Alivanis P. Lactic acidosis after concomitant treatment with metformin and tenofovir in a patient with HIV infection. J Ren Care. 2011 Mar;37(1):25-9. doi: 10.1111/j.1755-6686.2011.00209.x. PMID 21288314
- [Background] Ortiz-Brizuela E, Perez-Patrigeon S, Recillas-Gispert C, Gomez-Perez FJ. Lactic Acidosis Complicating Metformin and Non-Nucleoside Reverse Transcriptase Inhibitor Combination Therapy: A Smoldering Threat in the Post-HAART Era. Rev Invest Clin. 2015 Jul-Aug;67(4):273-4. PMID 26426594
- [Background] Ledvina M, Bartos F, Hroch M. Formation of hydroxyproline-containing proteins by fibroblasts in tissue culture (chick embryo fibroblasts-L-cells- 14 C proline-labelling). Folia Biol (Praha). 1972;18(5):327-30. No abstract available. PMID 4636755
- [Background] Naccarato M, Yoong D, Fong IW. Dolutegravir and metformin: a case of hyperlactatemia. AIDS. 2017 Sep 24;31(15):2176-2177. doi: 10.1097/QAD.0000000000001617. No abstract available. PMID 28906282
- [Background] Cho SK, Yoon JS, Lee MG, Lee DH, Lim LA, Park K, Park MS, Chung JY. Rifampin enhances the glucose-lowering effect of metformin and increases OCT1 mRNA levels in healthy participants. Clin Pharmacol Ther. 2011 Mar;89(3):416-21. doi: 10.1038/clpt.2010.266. Epub 2011 Jan 26. PMID 21270793
- [Background] Roberts C, Nylander AE, Jayaramachandran S. Orbital cellulitis complicating isolated unilateral sphenoidal sinusitis: importance of the CT scan. Br J Ophthalmol. 1989 Sep;73(9):769-70. doi: 10.1136/bjo.73.9.769. PMID 2804035
- [Background] Doyle MA, Singer J, Lee T, Muir M, Cooper C. Improving treatment and liver fibrosis outcomes with metformin in HCV-HIV co-infected and HCV mono-infected patients with insulin resistance: study protocol for a randomized controlled trial. Trials. 2016 Jul 20;17(1):331. doi: 10.1186/s13063-016-1454-6. PMID 27439433
- [Background] Cameron AR, Morrison VL, Levin D, Mohan M, Forteath C, Beall C, McNeilly AD, Balfour DJ, Savinko T, Wong AK, Viollet B, Sakamoto K, Fagerholm SC, Foretz M, Lang CC, Rena G. Anti-Inflammatory Effects of Metformin Irrespective of Diabetes Status. Circ Res. 2016 Aug 19;119(5):652-65. doi: 10.1161/CIRCRESAHA.116.308445. Epub 2016 Jul 14. PMID 27418629
- [Background] Lazarus B, Wu A, Shin JI, Sang Y, Alexander GC, Secora A, Inker LA, Coresh J, Chang AR, Grams ME. Association of Metformin Use With Risk of Lactic Acidosis Across the Range of Kidney Function: A Community-Based Cohort Study. JAMA Intern Med. 2018 Jul 1;178(7):903-910. doi: 10.1001/jamainternmed.2018.0292. PMID 29868840
- [Background] Moyo S, Bussmann H, Mangwendeza P, Dusara P, Gaolathe T, Mine M, Musonda R, van Widenfelt E, Novitsky V, Makhema J, Marlink RG, Essex M, Wester CW. Validation of A Point-of-Care Lactate Device For Screening At-Risk Adults Receiving Combination Antiretroviral Therapy In Botswana. J Antivir Antiretrovir. 2011 Oct;3(4):45-48. doi: 10.4172/jaa.1000034. Epub 2011 Sep 20. PMID 23087782